CLINICAL TRIAL: NCT07240298
Title: Comparison of Triglyceride-Glucose Index and Atherogenic Indices Between Patients With Lipedema and Obese Controls: A Cross-Sectional Study
Brief Title: Comparison of Triglyceride-Glucose Index and Atherogenic Indices Between Patients With Lipedema and Obese Controls
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Fatma Nur Kesiktaş, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: istftreah1
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Lipedema
MeSH Terms: conditions — Lipedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lipedema group: Obese patients with lipedema
  Interventions: Other: No intervention
- Control group: Obese patients without lipedema
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Women aged 18-75 years with a clinical diagnosis of lipedema and an obese control group will be included in the study. Sociodemographic and clinical data (age, height, weight, medications, etc.) of the participants will be recorded. For laboratory evaluation, fasting blood test results obtained within the last three months (including fasting glucose, total cholesterol, LDL-cholesterol, HDL-cholesterol, and triglycerides) will be used. Based on these parameters, metabolic and atherogenic risk indicators such as the Triglyceride-Glucose Index (TyG), TyG-BMI, Atherogenic Index of Plasma (AIP), Atherogenic Coefficient (AC), Castelli Risk Index I (CRI-I), and Castelli Risk Index II (CRI-II) will be calculated. No additional biochemical tests will be collected from participants; analyses will be performed using existing laboratory results.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with lipedema
* Obese control group with BMI ≥30 kg/m² who do not meet lipedema criteria
* Aged between 18 and 75 years
* Availability of fasting lipid profile and fasting glucose tests within the past 3 months
* Provided voluntary informed consent

Exclusion Criteria:

* Use of medications that routinely affect lipid or glucose metabolism: statins, fibrates, niacin, ezetimibe, high-dose omega-3 supplements, GLP-1 receptor agonists, SGLT2 inhibitors, or systemic corticosteroids (regular use within the past 3 months)
* Presence of rheumatologic diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus) or active malignancy
* Neurological disorders (e.g., polyneuropathy, multiple sclerosis, history of stroke)
* Pregnancy or lactation
* History of lower extremity surgery or major trauma within the past 6 months
* Received injection therapy or physical therapy for the lower extremities within the past 6 months
* Active infection or dermatological disease affecting the lower extremities
* History of significant venous insufficiency or acute deep vein thrombosis (DVT)
* Alcohol or substance abuse
* Smoking

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: obese patients with and without lipedema
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2025-10-10 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Triglyceride-Glucose Index (TyG): | Baseline
  The TyG index will be calculated as ln [fasting triglycerides (mg/dL) × fasting glucose (mg/dL) / 2]. It serves as a surrogate marker for insulin resistance. Higher values indicate greater metabolic risk.

SECONDARY OUTCOMES:
TyG-BMI | Baseline
  Calculated by multiplying the TyG index by body mass index (BMI). Higher values indicate increased insulin resistance and metabolic risk.
Atherogenic Index of Plasma (AIP): | Baseline
  Calculated as log (triglycerides / HDL-cholesterol). Higher AIP values reflect greater atherogenic risk.
Atherogenic Coefficient (AC): | Baseline
  Calculated as (total cholesterol - HDL-cholesterol) / HDL-cholesterol. Higher scores indicate higher atherogenic potential.
Castelli Risk Index I (CRI-I): | Baseline
  Calculated as total cholesterol / HDL-cholesterol. Higher values indicate increased cardiovascular risk.
Castelli Risk Index II (CRI-II): | Baseline
  Calculated as LDL-cholesterol / HDL-cholesterol. Higher scores represent greater atherogenic risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)